CLINICAL TRIAL: NCT06758713
Title: Safety and Efficacy of Fourth-Generation CAR-T in the Treatment of Hematologic Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The Third Affiliated Hospital of Southern Medical University (Other Government)
Responsible Party: Principal Investigator, Yan Yi, MD., The Third Affiliated Hospital of Southern Medical University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-Lunli-020; 2024-Lunli-020 (Other: The clinical Trial Ethics Committee)
Record Dates: First submitted 2024-12-27; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-07

CONDITIONS: Multiple Myeloma; B-cell Lymphoma; Hematological Malignancy
Keywords: Multiple myeloma; B-cell lymphoma; Hematological malignancy; CAR-T; Safety; Efficacy
MeSH Terms: conditions — Multiple Myeloma; Lymphoma, B-Cell; Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Phase 1:Low dose group (Experimental): Infusion of CAR T-cells by single dose of 0.5×10^6 CAR-T cells/kg
  Interventions: Biological: CAR-T
- Phase 1: Medium dose group (Experimental): Infusion of CAR T-cells by single dose of 1.5×10^6 CAR-T cells/kg
  Interventions: Biological: CAR-T
- Phase 1: High dose group (Experimental): Infusion of CAR T-cells by single dose of 5.0×10^6 CAR-T cells/kg
  Interventions: Biological: CAR-T
- Phase 2a: RP2D (Experimental): After all subjects in the Phase 1 dose-escalation study completed DLT observation, RP2D was determined based on the analysis results for the phase 2a expansion study.
  Interventions: Biological: CAR-T

INTERVENTIONS:
Biological: CAR-T — CAR T-cell therapy involves autologous chimeric antigen receptor T-cells, capable of targeting human B cell maturation antigen (BCMA) ,CD19 or CD-7 etc. target molecules of other hematologic malignancies.

SUMMARY:
This is a single center, open-label, dose-escalation/expansion clinical study to evaluate the safety and effectiveness of Fourth-Generation CAR-T, and determine the recommended dose of the CAR T-cells for patients with Multiple Myeloma，B-cell lymphoma and other hematologic malignancies.

DETAILED DESCRIPTION:
This is a single center, open-label, dose-escalation/expansion clinical study to evaluate the safety and efficacy of Fourth-Generation CAR-T in the Treatment of Multiple Myeloma，B-cell lymphoma and other hematologic malignancies.. -Prior to Fourth-Generation CAR-T cells infusion, subjects will receive lymphodepleting therapy with fludarabine and cyclophosphamide. After infusion, the investigators will observe the characteristics of dose limited toxicity (DLT), and determine the maximum tolerable agent MTD and RP2D were confirmed. To provide basis for the dosage and treatment plan of cell products in follow-up clinical trials. Meanwhile, subjects will be followed for side effects and effect of the CAR-T.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to be enrolled:

1. Voluntarily participate in this clinical study and sign the informed consent form; 2. 18 to 75 years old (including cut-off value), Male and female;; 3. Expected survival of at least 3 months; 4.1 CD19-positive B lymphocyte-derived hematologic malignancies; 4.2 Multiple myeloma patients; 4.3 Non-B cell-derived hematologic malignancies patients with CD7 or other target molecules; 5. The clinical trial values during the screening period meet the following criteria:

1. White blood cell count ≥ 3.0 × 10e9/L; Absolute neutrophil ≥ 1.0 × 10e9/L; Lymphocyte count ≥ 0.5 × 10e9/L. (The growth factor support is allowed, but growth factor must not have been received within 7 days prior to laboratory testing);
2. Platelet count ≥ 50 × 10e9/L (No blood transfusion support within 7 days prior to laboratory tests.); Note: Patients with leukemia, multiple myeloma, and lymphoma are not subject to the above blood picture requirements;
3. Biochemical indicators Serum total bilirubin (TBIL) ≤ 2.5 ULN, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 ULN, or 5 ULN if liver dysfunction is primarily due to tumor invasion); 6. Cardiac function: Subjects must have good hemodynamic stability, left ventricular ejection fraction (LVEF) ≥ 55%; 7. Lung condition: Subjects are not serious infections such as severe pneumonia; 8. ECOG activity status score: 0-2 points; 9. Female subjects must use effective contraception (such as oral prescription contraceptives, injectable contraceptives, intrauterine devices, double blockade, contraceptive patches, male partner sterilization) throughout the study period; Must have a negative serum or urine pregnancy test result at screening and throughout the study.

Exclusion Criteria:

Any one of the following conditions cannot be selected as a subject:

1. Having received CAR-T therapy targeting the same molecule;
2. Having received other immunotargeted therapy targeting the same molecules;
3. Pregnant or lactating women;
4. Subjects who have previously suffered from other malignancies, with the following exceptions:

   1. Having received curative therapy, and no known active disease in the ≥ 3 years prior to the enrollment;
   2. Non melanoma skin cancer subjects who have completed sufficient treatment and no evidence of thecurrent disease;
5. Subjects with a severe mental disorder;
6. Subjects with active autoimmune disease requiring immunotherapy;
7. Having received allogeneic hematopoietic stem cell transplantation;
8. Subjects with significant cardiovascular diseasesa.uncontrolled or symptomatic arrhythmias, congestive heart failure, or any heart disease with cardiac function grade 3 or grade 4 (according to the functional classification method of the New York Heart Association NYHA); b. Myocardial infarction or coronary artery bypass grafting within 6 months prior to screening); c. Clinically significant history of ventricular arrhythmia or unexplained syncope (non vaso-vagal or not due to dehydration);
9. Subjects with active infectious disease including positive Hepatitis B surface antigen (HBsAg) or Hepatitis B core antibody (HBcAb) and peripheral blood Hepatitis B virus(HBV) DNA titer is ≥500IU/mL, hepatitis C virus (HCV) antibody positive and peripheral blood HCV RNA positive, human immunodeficiency virus(HIV) antibody positive, syphilis primary screening antibody positive, active pulmonary tuberculosis; or with any significant infection requiring high-grade antibiotics Event;
10. Subjects with dysfunction of important organssuch as organ function in the following abnormalities:

    1. Serum AST or ALT > 2.5×ULN, or > 5ULN if liver function is predominantly due to tumor invasion; TBIL > 2.5 × ULN, unless the subject is Gilbert's syndrome;
    2. Serum creatinine>2.5mg/dl;
    3. Partial prothrombin time or activated partial thromboplastin time or international normalized ratio > 1.5×ULN in the absence of anticoagulant therapy;
11. Participation in other clinical studies or prior treatment with any gene therapy product in the past three months;
12. Subjects with uncontrolled diabetes mellitus (glycosylated hemoglobin HbAlc >8% at screening);13. Highly allergic constitution or history of severe allergies, and having contraindications to cyclophosphamide or fludarabine;

14. Feasibility assessment screening demonstrated <10% transfection of targeted lymphocytes or underamplification under CD3 / CD28 costimulation (<5-fold); 15. Subjects who are considered unsuitable to participate in this trial by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with dose-limiting toxicity (DLT) | Within 30 days of receiving CAR T-cells transfusion therapy
  For DLT evaluation, severity (grade) is classified according to common terminology criteria for adverse events version 4.03 (CTCAE v4.03).
Maximum Tolerated Dose (MTD) | Within 30 days of receiving CAR T-cells transfusion therapy
  At least 6 subjects in the MTD dose group must complete the DLT assessment.
Adverse Event | Minimum 2 years after CAR T-cells infusion (Day 1)
  Safety will be assessed by adverse events (AEs), which include clinically significant abnormalities identified during medical tests (e.g. laboratory tests, electrocardiogram, imaging examinations or physical examinations). AEs will be coded by Medical Dictionary for Regulatory Activities (MeDRA) and their severity will be graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE, version 4.03).
Recommended Phase 2 Dose (RP2D) | Through study completion, an average of 1 year
  To determine after all subjects in the Phase 1 dose-escalation study completed DLT observation
Objective response rate (ORR) | Through study completion, an average of 2 years
  The definition of ORR is the proportion of subjects achieving sCR, CR, VGPR, or PR confirmed by efficacy reassessment after a minimum interval of three months. ORR is calculated as (sCR+CR+VGPR+PR) divided by the total number of cases of Multiple Myeloma, or (CR+PR) divided by the total number of cases of B-cell lymphoma and other hematologic malignancies, multiplied by 100%.

SECONDARY OUTCOMES:
Stringent complete response rate (sCRR) | Through study completion, an average of 2 years
  The definition of sCRR is the proportion of subjects achieving sCR confirmed by efficacy re-assessment after a minimum interval of three months. Efficacy assessment for multiple myeloma only.
Progression-free Survival (PFS) | Through study completion, an average of 2 years
  The time interval from the first administration of the investigational drug to the first observation of disease progression is calculated, considering the date of entry for patients who died for reasons other than disease progression before progression occurred.
Overall Survival (OS) | Through study completion, an average of 2 years
  OS is the time from the start of cell infusion to the death of the subject.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Yi, MD., Study Director
Locations (1):
- The Third Affiliated Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roddie C, Dias J, O'Reilly MA, Abbasian M, Cadinanos-Garai A, Vispute K, Bosshard-Carter L, Mitsikakou M, Mehra V, Roddy H, Hartley JA, Spanswick V, Lowe H, Popova B, Clifton-Hadley L, Wheeler G, Olejnik J, Bloor A, Irvine D, Wood L, Marzolini MAV, Domning S, Farzaneh F, Lowdell MW, Linch DC, Pule MA, Peggs KS. Durable Responses and Low Toxicity After Fast Off-Rate CD19 Chimeric Antigen Receptor-T Therapy in Adults With Relapsed or Refractory B-Cell Acute Lymphoblastic Leukemia. J Clin Oncol. 2021 Oct 20;39(30):3352-3363. doi: 10.1200/JCO.21.00917. Epub 2021 Aug 31. PMID 34464155
- [Background] Sang W, Wang X, Geng H, Li T, Li D, Zhang B, Zhou Y, Song X, Sun C, Yan D, Li D, Li Z, Li C, Xu K. Anti-PD-1 Therapy Enhances the Efficacy of CD30-Directed Chimeric Antigen Receptor T Cell Therapy in Patients With Relapsed/Refractory CD30+ Lymphoma. Front Immunol. 2022 Apr 1;13:858021. doi: 10.3389/fimmu.2022.858021. eCollection 2022. PMID 35432352
- [Background] Du J, Wei R, Jiang S, Jiang H, Li L, Qiang W, He H, Shi L, Ma Q, Yu K, Zhang X, Ding H, Sun X, Xiang F, Zhu L, Cheng Z, Fu W. CAR-T cell therapy targeting B cell maturation antigen is effective for relapsed/refractory multiple myeloma, including cases with poor performance status. Am J Hematol. 2022 Jul;97(7):933-941. doi: 10.1002/ajh.26583. Epub 2022 May 5. PMID 35488407
- [Background] Yang J, He J, Zhang X, Li J, Wang Z, Zhang Y, Qiu L, Wu Q, Sun Z, Ye X, Yin W, Cao W, Shen L, Sersch M, Lu P. Next-day manufacture of a novel anti-CD19 CAR-T therapy for B-cell acute lymphoblastic leukemia: first-in-human clinical study. Blood Cancer J. 2022 Jul 7;12(7):104. doi: 10.1038/s41408-022-00694-6. PMID 35798714
- [Background] Qu C, Zou R, Wang P, Zhu Q, Kang L, Ping N, Xia F, Liu H, Kong D, Yu L, Wu D, Jin Z. Decitabine-primed tandem CD19/CD22 CAR-T therapy in relapsed/refractory diffuse large B-cell lymphoma patients. Front Immunol. 2022 Aug 17;13:969660. doi: 10.3389/fimmu.2022.969660. eCollection 2022. PMID 36059523
- [Background] Ying Z, Xie Y, Zheng W, Liu W, Lin N, Tu M, Wang X, Ping L, Deng L, Zhang C, Wu M, Feng F, Du T, Tang Y, Su F, Guo Z, Li J, Song Y, Zhu J. Efficacy and safety of relmacabtagene autoleucel, an anti-CD19 chimeric antigen receptor T cell, in relapsed/refractory B-cell non-Hodgkin's lymphoma: 2-year results of a phase 1 trial. Bone Marrow Transplant. 2023 Mar;58(3):288-294. doi: 10.1038/s41409-022-01888-z. Epub 2022 Dec 7. PMID 36477110
- [Background] Liang EC, Albittar A, Huang JJ, Hirayama AV, Kimble EL, Portuguese AJ, Chapuis A, Shadman M, Till BG, Cassaday RD, Milano F, Kiem HP, Riddell SR, Turtle CJ, Maloney DG, Gauthier J. Factors associated with long-term outcomes of CD19 CAR T-cell therapy for relapsed/refractory CLL. Blood Adv. 2023 Nov 28;7(22):6990-7005. doi: 10.1182/bloodadvances.2023011399. PMID 37774014
- [Background] Minson A, Hamad N, Cheah CY, Tam C, Blombery P, Westerman D, Ritchie D, Morgan H, Holzwart N, Lade S, Anderson MA, Khot A, Seymour JF, Robertson M, Caldwell I, Ryland G, Saghebi J, Sabahi Z, Xie J, Koldej R, Dickinson M. CAR T cells and time-limited ibrutinib as treatment for relapsed/refractory mantle cell lymphoma: the phase 2 TARMAC study. Blood. 2024 Feb 22;143(8):673-684. doi: 10.1182/blood.2023021306. PMID 37883795